CLINICAL TRIAL: NCT00529672
Title: Randomized Single Center Comparative Study of the Treatment of Insufficient Greater Saphenous Vein: Surgery vs Ultrasound Guided Sclerotherapy With Foam and Endovenous Laser Therapy
Brief Title: Surgery or Noninvasive Therapy for Varicose Veins
Acronym: Magna
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Dr. TEC Nijsten, Erasmus MC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-325
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Varicose Vein
Keywords: endovenous laser therapy; sclerotherapy; crossectomy and stripping; surgery; treatment; varicose veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Surgery: crossectomy plus short stripping
  Interventions: Procedure: crossectomy and short stripping
- 2 (Active Comparator): ultrasound guided sclerotherapy with foam (3% polidocanol)
  Interventions: Procedure: ultrasound guided sclerotherapy with foam
- 3 (Active Comparator): Endovenous laser therapy (940 nm, about 70 J/cm)
  Interventions: Procedure: endovenous laser therapy

INTERVENTIONS:
Procedure: crossectomy and short stripping — under spinal or complete anaesthesia
  Arms: 1
Procedure: ultrasound guided sclerotherapy with foam — 1 part 3% polidocanol mixed with 3 parts of air. Between 3cc - 12 cc per varicose vein>
  Arms: 2
Procedure: endovenous laser therapy — 940 nm Diode laser. About 70 J/cm will be administered. Disposables from Angiocare (registered) will be used.
  Arms: 3

SUMMARY:
For more than 100 years, surgery has been the standard of care of varicose veins of the legs. The down side of surgery is that it requires anesthesia, leaves scars, and has a relatively high recurrence rate in the long term (up to 40%). In the last decade, several new techniques have become available but they have not yet been compared to surgery. This trail will evaluate the effectiveness, patients' perspective and cost effectiveness of surgery and non-invasive techniques such as ultrasound guided sclerotherapy with foam and endovenous laser therapy.

DETAILED DESCRIPTION:
Inclusion criteria:

* Ultrasound confirmed GSV insufficiency (reflux time >0.5 second and vein diameter ≥0.5 cm)
* non-treated GSV varicosis
* CEAP -classification > C2 and As2
* >18 years old
* Informed consent.

Exclusion criteria:

* Acute venous thrombosis / phlebitis
* Absence of deep venous system
* Vascular syndromes
* Post-thrombotic syndrome of occlusive type
* Contra-indications for surgery
* use of anticoagulants

Primary outcomes:

1. anatomical success using US (absence of GSV or flow) (at 3 months, 1 and 5 year)

Secondary outcomes:

1. treatment induced adverse events and complications (after 3 months)
2. patient reported outcomes (HRQOL and treatment satisfaction)(after 3 months)
3. cost effectiveness analyses (after 1 and 5 years)

Included patients: total of 240 (80 per arm)

Study start: May 2007 (recruitment ongoing) Study completion: May 2011

Follow up after 3 months, 1, 2, 3, 4 and 5 years

Location: department of dermatology, Erasmus MC, Rotterdam, The Netherlands

Principle investigators: M. Kockaert, T. Nijsten & M. Neumann

Publications:

Rasmussen LH, Bjoern L, Lawaetz M, Blemings A, Lawaetz B, Eklof B. Randomized trial comparing endovenous laser ablation of the great saphenous vein with high ligation and stripping in patients with varicose veins: short-term results. J Vasc Surg. 2007 Aug;46(2):308-15. Epub 2007 Jun 27.

Sharif MA, Lau LL, Lee B, Hannon RJ, Soong CV. Role of endovenous laser treatment in the management of chronic venous insufficiency. Ann Vasc Surg. 2007 Sep;21(5):551-5.

Mundy L, Merlin TL, Fitridge RA, Hiller JE. Systematic review of endovenous laser treatment for varicose veins. Br J Surg. 2005 Oct;92(10):1189-94.

Jia X, Mowatt G, Burr JM, Cassar K, Cook J, Fraser C.Systematic review of foam sclerotherapy for varicose veins. Br J Surg. 2007 Aug;94(8):925-36.

Subramonia S, Lees TA.The treatment of varicose veins.Ann R Coll Surg Engl. 2007 Mar;89(2):96-100.

Bohler K. Varicose veins: disfigurement or disease? Herz. 2007 Feb;32(1):18-25.

Bamigboye AA, Smyth R. Interventions for varicose veins and leg oedema in pregnancy. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD001066.

van den Bos R, Arends L, Kockaert M, Neumann M, Nijsten T. New endovenous therapies of truncal varicosities are more effective than surgical stripping and sclerotherapy: meta-analysis and meta-regression. Lancet, Submitted

ELIGIBILITY:
Inclusion Criteria:

* primary insufficient GSV confirmed by US: reflux>0.5 sec and diameter>0.5cm.
* non-treated insufficient GSV
* >18 years
* informed consent

Exclusion Criteria:

* acute thrombosis or phlebitis
* absence of deep venous system
* vascular syndromes
* use of anticoagulants
* contraindications surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2007-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
anatomical success rate (absence or obliteration of GSV on US examination) | 3 months, 1 and 5 years

SECONDARY OUTCOMES:
treatment related adverse events and complications | 3 months, 1 and 5 years
patient reported outcomes (HRQOL and treatment satisfaction) | 3 months, 1 and 5 years
cost effectiveness analysis | 3 months, 1 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Martino Neumann, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC dermatology, Rotterdam, Netherlands

REFERENCES:
- [Derived] van der Velden SK, Biemans AA, De Maeseneer MG, Kockaert MA, Cuypers PW, Hollestein LM, Neumann HA, Nijsten T, van den Bos RR. Five-year results of a randomized clinical trial of conventional surgery, endovenous laser ablation and ultrasound-guided foam sclerotherapy in patients with great saphenous varicose veins. Br J Surg. 2015 Sep;102(10):1184-94. doi: 10.1002/bjs.9867. Epub 2015 Jul 1. PMID 26132315
- [Derived] Biemans AA, Kockaert M, Akkersdijk GP, van den Bos RR, de Maeseneer MG, Cuypers P, Stijnen T, Neumann MH, Nijsten T. Comparing endovenous laser ablation, foam sclerotherapy, and conventional surgery for great saphenous varicose veins. J Vasc Surg. 2013 Sep;58(3):727-34.e1. doi: 10.1016/j.jvs.2012.12.074. Epub 2013 Jun 13. PMID 23769603